CLINICAL TRIAL: NCT06951035
Title: ETUDE DE L'AMELIORATION DU CONTROLE DES INTERFACES CERVEAU-MACHINE PAR LA CONNECTIVITE FONCTIONNELLE ET LA STIMULATION MAGNETIQUE TRANSCRANIENNE REPETEE DANS LA REEDUCATION MOTRICE DU MEMBRE SUPERIEUR APRES UN ACCIDENT VASCULAIRE CHRONIQUE
Brief Title: Impact of rTMS on BCI Control in Upper Limb Motor Rehabilitation of Patients With Chronic Stroke
Acronym: BCINET
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C23-46; 2024-A00230- 47 (Registry Identifier: IDRCB)
Record Dates: First submitted 2025-04-15; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Chonic Stroke Patients With Motor Impairment of Upper Limb
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Randomised Mutliple Baseline SCED.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- rTMS-free group (No Intervention): Chronic stroke patients with motor deficit of upper limb
- Contralesional Inhibitory stimulation of the M1 cortex. (Experimental): The probe will be placed on the healthy motor cortex at the Extensor Carpi Radialis " hotspot " level.
  Performed on 15 participants (5 participants per group)
  * Group A : chronic stroke with severe upper limb motor deficit (UE-FMA score ≤ 31)
  * Group B : chronic stroke with mild upper limb motor deficit (UE-FMA score > 31)
  * Group C : chronic stroke with upper limb motor deficit with hemineglect
  Interventions: Device: Repetitive transcranial magnetic stimulation (rTMS)
- Ipsilesional excitatory stimulation of the M1 cortex. (Experimental): The probe will be placed on the injured motor cortex at the Extensor Carpi Radialis " hotspot " level.
  Performed on 15 participants (5 participants per group)
  * Group A : chronic stroke with severe upper limb motor deficit (UE-FMA score ≤ 31)
  * Group B : chronic stroke with mild upper limb motor deficit (UE-FMA score > 31)
  * Group C : chronic stroke with upper limb motor deficit with hemineglect
  Interventions: Device: Repetitive transcranial magnetic stimulation (rTMS)
- Personalized exitatory stimulation according to structural connectivity. (Experimental): The probe will be placed at the stimulation site identified by control theory. Performed on 15 participants (5 participants per group)
  * Group A : chronic stroke with severe upper limb motor deficit (UE-FMA score ≤ 31)
  * Group B : chronic stroke with mild upper limb motor deficit (UE-FMA score > 31)
  * Group C : chronic stroke with upper limb motor deficit with hemineglect
  Interventions: Device: Repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation (rTMS) — The repeated stimulations will be carried out using an eight-part probe detected by the infrared camera ("eight shaped tracked coil"), connected to a Rapid 2 stimulator (Magstim Company, Whitland, UK). The stimulation will be performed manually or with robotic assistance using TMS-Robot (Axilum Robotics, SCHILTIGHEIM, France)
  Arms: Contralesional Inhibitory stimulation of the M1 cortex.; Ipsilesional excitatory stimulation of the M1 cortex.; Personalized exitatory stimulation according to structural connectivity.

SUMMARY:
Cerebrovascular accidents (strokes) are a major public health issue. Stroke is the 3rd leading cause of death and the leading cause of disability and loss of autonomy. In France, there are currently 130,000 new cases per year, and the aging of the population will lead to an increase in this number over the next few years. Among post-stroke impairments, motor deficit of the upper limb is the most common disability, affecting 73-88% of first-time stroke patients and 55-75% of chronic patients. Associated deficits can complicate rehabilitation management and affect recovery. The clinical profile of patients with motor deficits is therefore varied and complex, requiring an individualized approach. At present, only physiotherapy is recommended, with modest results.

Repeated transcranial magnetic stimulation is a therapy that can improve motor recovery, but currently has a low level of evidence according to the HAS (French Hight Health Authority), notably because of variability in efficacy due to heterogeneity in the clinical profile of patients. Nevertheless, it is still recommended for the recovery of cognitive functions, but also for resistant depression, and could be used to stimulate motor imagery (MI). MI training also has the advantage of stimulating the motor network. Difficult to achieve for a number of patients, the use of rTMS could facilitate this cognitive task and, in particular, provide better access to brain-computer interfaces (BCI). Indeed, among the innovative rehabilitation therapies, BCIs have emerged as the most promising. By translating brain activity during a cognitive task into a command such as electrical muscle stimulation, BCIs would restore the damaged motor network and induce motor recovery. The main obstacle to their widespread use in clinical practice is their lack of reliability, as almost 30% of patients are unable to control them correctly, either because of difficulty in performing the MI task, or because of difficulty in identifying a universal brain signature.

The BCINET project aims to improve the reliability of BCIs in two ways: by improving detection of the motor imagination task using new brain signatures, and through cognitive facilitation using rTMS.

1. - Using the dynamic communication of different brain areas during the MI task (or functional connectivity), we can identify patient-specific signatures. Studies of functional connectivity in healthy subjects performing an MI task without associated BCI have shown the interest of certain measures such as node degree or clustering coefficient. To find out whether functional connectivity parameters can be used in BCI algorithms, we will evaluate their effectiveness on an initial group of 5 patients to define their performance in discriminating the MI task and to determine their evolution over time in the absence of brain stimulation in stroke patients. Their initial study will also enable us to identify their evolution when TMS stimulation is applied.
2. - Cerebral magnetic stimulation could facilitate the MI task and enable better BCI rehabilitation for a number of patients. Two studies using either an inhibitory or excitatory stimulation protocol showed an improvement in spectral power signal and better discrimination of the MI task. However, the results were acquired using a single pre- and post-therapy measurement, and did not take into account behavioral variability in the use of BCIs or variability in TMS response according to patient profile. Therefore, in order to identify whether rTMS would improve BCI control, we would perform 9 Single-Case Experimental Design (SCED) studies in multiple baselines on a group of 5 patients according to 3 clinical profiles and 3 rTMS stimulation strategies. SCEDs are suitable experimental models for heterogeneous populations, particularly when the intervention presents some inter-individual variability in efficacy. They have the advantage of being able to demonstrate, on an individual scale, the effectiveness of the intervention on a small group of patients. Replication of the SCED allows us to increase the external validity of the intervention on sub-groups of patients (clinical severity, presence of associated hemineglect) and to study modifications in the interventional strategy (stimulation frequency, stimulation site).

ELIGIBILITY:
Inclusion Criteria:

* Single Stroke older than 6 months
* Distal motor deficit of the upper limb (UE-FMA score < 53) with visible extension of the fingers (Medical Research Council (mRC) score ≥ 2)
* Right-handed
* Between 18 and 85 years of age
* Having given their written consent

Exclusion Criteria:

* Patient under tutorship or guardianship, under safeguard of justice, deprived of liberty, pregnant or breast feeding women
* Life-threatening pathologies or compromising follow-up during the study period
* Trouble of understanding : score below 12/15 in the Boston Diagnostic Aphasia Examination (BDAE) order execution test
* Fixed spasticity of finger or carpal flexors (mAS score = 4) or botulinum toxin injection less than 12 weeks old in the forearm or hand
* History of degenarative neurological pathology or craniectomy
* Deficient upper limb skin lesion preventing use of mucle stimulation
* Skin lesion of the scalp preventing EEG placement
* Participation in biomedical therapeutic research that may affect the recovery of the deficient hand during the study
* Patient who has previously participated in a therapeutic study rTMS (excluding single shock) or a BCI
* Patient who does not wish to be informed of a brain abnormality discovered accidentally on MRI

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Measuring primary BCI performance | 6 weeks, 18 weeks
  Accuracy was choosen, which correspond to the percentage of correct detection of mental tasks (either MI or rest) on all tasks performed during the session.

SECONDARY OUTCOMES:
Measuring secondary BCI performance by using the sensitivity indicator " recall " | Up to 20 weeks
  Sensitivity is the proportion of correct IM task detections out of all real IM tasks
Measuring secondary BCI performance by using the positive predictive value " precision " | Up to 20 weeks
  The positive predictive value is the proportion of correct MI detections out of all tasks detected by algorithm
Measuring secondary BCI performance by using the Run-Wise Cross-Validation method | Up to 20 weeks
  To reduce the the intersessional variabilityy in accurnc, we use the Run-Wise Cross-Validation (RWCV CA) method will be used.
Assessment of the motor function using the Fugl-Meyer upper limb motor subscale (UE-FMA) | Inclusion visit, 6 weeks
  Rough assessment of dexterity during goal directed movements
Assessment of the motor function using Box and Block Test (BBT) | Up to 20 weeks
  Rough assessment of dexterity during goal directed movements
Assessment of the motor function using the Grip and Pinch force | Up to 20 weeks
  Pure evaluation of the finger flexion force using dynamometer
Evaluation of spasticity | Inclusion visit, 6 weeks
  Will be assessed and monitored using the modified Ashworth scale (mAs score)
Hemineglet assessment by text reading test | Up to 20 weeks
  A text reading test in which the number of words correctly read in one minute and the percentage of words omitted will be counted
Hemineglet assessment by line bissection test | Up to 20 weeks
  The measurement of the center deviation will be quantified
Analysis of spectral power | Up to 20 weeks
  Measurement of the power of electrical signal produced by the brain depending on frequency
Phase-Amplitude Coupling (PAC) analysis | Up to 20 weeks
  By analysing the phase-amplitude relationships of different frequency bands in the EEG signal
Quantification of the functional connectivity (FC) | 2 minutes before starting rTMS stimulation
  To quantify this communication, we will use a correlation matrix constructed by calculating the coefficients of spectral coherence between all of EEG channels pairs
Measurement of cortical excitability (Motor Evoked Potentials) | Inclusion visit, 6 weeks, 18 weeks
  Assessment of the amplitude of MEPs per single shock TMS and representes the therapeutic target of rTMS

CONTACTS AND LOCATIONS:
Locations (1):
- Institut du Cerveau, Paris, France

IPD SHARING:
Plan to Share IPD: No